CLINICAL TRIAL: NCT06582758
Title: Brief (<10 Minute) Behavioral Interventions for Pain
Brief Title: Does Choice Improve the Pain Relief Derived From a Brief Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004916_MOD5065
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pain; Acute Pain
Keywords: mindfulness
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindful Pain Management (randomized) (Experimental): In the control mindful pain management intervention, participants will be randomized to listen to a four minute mindfulness intervention consisting of a 1-minute introduction to mindful pain management and a 3-minute mindfulness practice.
  Interventions: Behavioral: Mindful Pain Management
- Pain Psychoeducation (randomized) (Active Comparator): In the pain psychoeducation intervention, participants will be randomized to listen to a four-minute recording about different pain management strategies (e.g., ice, rest) and accessible resources to promote overall well-being.
  Interventions: Behavioral: Pain Psychoeducation
- Choice: Mindful Pain Management (Experimental): In the choice mindful pain management intervention, participants will choose to listen to a four minute mindfulness intervention consisting of a 1-minute introduction to mindful pain management and a 3-minute mindfulness practice.
  Interventions: Behavioral: Mindful Pain Management
- Choice: Pain Psychoeducation (Active Comparator): In the choice pain psychoeducation intervention, participants will choose to listen to a four-minute recording about different pain management strategies (e.g., ice, rest) and accessible resources to promote overall well-being.
  Interventions: Behavioral: Pain Psychoeducation

INTERVENTIONS:
Behavioral: Pain Psychoeducation — In the pain psychoeducation intervention, participants will be provided a four-minute recording about different pain management strategies (e.g., ice, rest) and accessible resources to promote overall well-being.
  Arms: Choice: Pain Psychoeducation; Pain Psychoeducation (randomized)
Behavioral: Mindful Pain Management — In the mindful pain management intervention, participants will listen to a four minute mindfulness intervention consisting of a 1-minute introduction to mindful pain management and a 3-minute mindfulness practice.
  Arms: Choice: Mindful Pain Management; Mindful Pain Management (randomized)

SUMMARY:
This project is a single-site, four-arm, randomized controlled trial investigating whether providing patients in an orthopedic clinic waiting room the ability to choose which pain management intervention the receive impacts the degree of pain relief they experience.

DETAILED DESCRIPTION:
This project is a single-site, four-arm, randomized controlled trial investigating whether providing patients in an orthopedic clinic waiting room the ability to choose which pain management intervention the receive impacts the degree of pain relief they experience. Participants will be randomized to one of three conditions: 1) a 4-minute pain psychoeducation recording, 2) a 4-minute mindfulness recording, or 3) choice. In the choice condition, participants will be able to choose which recoding (i.e., pain psychoeducation or mindfulness) they would like to listen to.

ELIGIBILITY:
Inclusion Criteria:

* Receiving pain treatment at Tallahassee Orthopedic Center
* Understanding English instructions fluently
* Being 18 years of age or older

Exclusion Criteria:

* Unable to consent because of physical or mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 7 to 10-minute audio recording
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 7 to 10-minute audio recording
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.
Change in Anxiety Numeric Rating Scale | Immediately before to after 7 to 10-minute audio recording
  Change in anxiety from baseline will be assessed with the Generalized Anxiety Disorder 2-item. Scores range from 0 to 6, with higher scores reflecting greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No